CLINICAL TRIAL: NCT05151276
Title: Effectiveness of Mobile Phone-based Distance Video Education in Individuals With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Mobile Phone-based Video Education on Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Özlem Tekir, Assist.Prof.Dr., Balikesir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BAUN"OTEKİR-001
Record Dates: First submitted 2021-10-23; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; diabetes education; mobile phone-based; distance video education; randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): individuals with odd sequence numbers were assigned to the intervention group (n=46)
  Interventions: Behavioral: mobile phone-based distance video education group
- Control Group (No Intervention): those with even numbers to the control group (n=47).

INTERVENTIONS:
Behavioral: mobile phone-based distance video education group — Following the first interview, diabetes education videos created previously were sent to the mobile phones of the individuals in two episodes a week fashion. Video submission was completed in a total of four weeks. In the second interview, three months after the video submission had been completed, data collection forms were re-administered to the individuals, and blood analysis results were recorded.
  Arms: Intervention Group

SUMMARY:
This study aimed to examine the effect of mobile phone-based distance video education given to individuals with type 2 diabetes on metabolic variables and cognitive-social factors. This study is a randomized controlled trial.

DETAILED DESCRIPTION:
MATERIALS AND METHODS:

This study is a randomized controlled trial.

Participants:

The population of the study consisted of individuals with type 2 diabetes who presented to hospital diabetes outpatient clinic between July 2018 and January 2019, and the study sample, on the other hand, included a total of 100 individuals with type 2 diabetes who met the inclusion criteria and agreed to participate in the study. The study was completed with a total of 93 subjects, including 46 in the intervention group (n = 46) and 47 in the control group (n= 47). A Diagnosis and Follow-up Form for Individuals with Diabetes (socio-demographic characteristics, diabetes-related characteristics, metabolic values), which was prepared by the researcher in line with the literature, and the Turkish Multidimensional Diabetes Questionnaire (T-MDDQ) were used to collect the data.

Preparation and content of the education material:

The education material was based on four different guidelines, namely, educator's guidelines for adults with diabetes; the diagnosis, treatment, and follow-up guidelines for diabetes mellitus and its complications; diabetes diagnosis and treatment guidelines; and international education guidelines for diabetes health professionals. The diabetes education videos prepared and presented by the researcher in line with these resources were sent to the participants' smartphones in parts. The educational content consisted of 8 sections: what is diabetes? (basic concepts, symptoms, diagnostic criteria, importance), medical nutrition therapy in diabetes, exercise therapy in diabetes, medical treatment in diabetes, acute complications of diabetes, chronic complications of diabetes, foot problems in diabetes, life with diabetes, and diabetes management under special cases.

Data collection process:

The intervention group: In the first meeting, the individuals in the intervention group were informed about the video-based diabetes education and how they would get the videos, and data collection forms were administered. The blood analysis results (HbA1c, glucose, total cholesterol, HDL, LDL, triglyceride) taken on the same day during outpatient clinic follow-ups were recorded. After the administration of the forms, blood pressure, height, and weight measurements were made, and the first interview was completed. Following the first interview, diabetes education videos created previously were sent to the mobile phones of the individuals in two episodes a week fashion. Video submission was completed in a total of four weeks. In the second interview, three months after the video submission had been completed, data collection forms were re-administered to the individuals, and blood analysis results were recorded. The interview was completed after measuring their blood pressure and weight. During the period between the first and second interviews, the individuals continued to receive routine outpatient follow-ups.

The control group: In the first interview, the individuals with diabetes in the control group were given information about the study, and then data collection forms were administered. The blood analysis results (HbA1c, glucose, total cholesterol, HDL, LDL, triglyceride) taken on the same day during outpatient clinic follow-ups were recorded. The first interview was completed after blood pressure, height, and weight measurements were made. Later, individuals continued to receive routine outpatient follow-ups without any other procedures. In the second interview held three months later, data collection forms were re-administered, and blood analysis results, blood pressure, and weight measurements were recorded. At the end of the second interview, diabetes education videos were sent to the individuals in the control group, too, and they were provided with the same education.

Data analysis:

The statistical package for social science (SPSS) version 25.0 (IBM Corp. Armonk, NY) was used to analyze the data. P<.05 was accepted statistically significant. In descriptive statistics, mean, ± standard deviation, median, minimum and maximum values, and percentages were used, and in nonparametric tests, Mann-Whitney U, Pearson's chi-square, Fisher's exact test, McNemar's test, Wilcoxon signed ranks test, and Spearman's rho measurements were employed.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Type 2 diabetes mellitus for at least 6 months.
* Being between the ages of 18-65.
* Being on oral antidiabetic and/or insulin therapy.
* Having a mobile phone capable of receiving and playing video messages.
* Volunteering to participate in the study.
* Sensory losses such as hearing and speech that will prevent communication

Exclusion Criteria:

* Being under 18 years of age
* Not having a mobile phone capable of receiving and playing video messages
* Not willing to participate in the study
* Having sensory loss such as hearing and speaking that prevents communication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The Turkish Multidimensional Diabetes Questionnaire | pre-test (baseline), post-test (3 months follow-up)
  Change from baseline diabetes-related cognitive and social factors at 3 months. Responses were on a Likert-type scale (0-not at all significant).
  not, 100-very important) is marked. High school scores perceived self-efficacy and outcome indicates high expectations.

SECONDARY OUTCOMES:
HbA1C | pre-test (baseline), post-test (3 months follow-up)
  HbA1C-change from baseline HbA1C at 3 months
glucose | pre-test (baseline), post-test (3 months follow-up)
  glucose -change from baseline glucose at 3 months
total cholesterol | pre-test (baseline), post-test (3 months follow-up)
  total cholesterol -change from baseline total cholesterol at 3 months
HDL | pre-test (baseline), post-test (3 months follow-up)
  HDL -change from baseline HDL at 3 months
LDL | pre-test (baseline), post-test (3 months follow-up)
  LDL -change from baseline LDL at 3 months
triglyceride | pre-test (baseline), post-test (3 months follow-up)
  triglyceride -change from baseline triglyceride at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kamil Bayraktar, Principal Investigator — Balikesir University
Locations (1):
- Balıkesir University, Balıkesir, Altıeylül, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No